CLINICAL TRIAL: NCT03536156
Title: Closure of Implant Emergence Profile
Acronym: FPEI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0181; 2018-A01269-46 (Other: ID-RCB)
Record Dates: First submitted 2018-05-09; First posted 2018-05-24 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Dental Implant
Keywords: Dental implant; Implant Emergence Profile

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Four intra-oral optical impression taken successively — Four intra-oral optical impression images will be taken successively on a patient:
  Optical impressions are designed to record adjacent implant site teeth and peri-implant soft tissue PEI using an Optical Camera. The optical camera works like a camera and does not come into contact with the patient's mucous membranes or teeth. The images obtained are saved in STL format on an anonymized file.
  The 4 aligned surfaces thus obtained will be cut using a 3D image processing software. A fixed cylinder will extract the PEI from the 4 surfaces. The volume of these 4 PEIs at T0 min, T30 sec, T2 min and T5 min will be calculated using a software

SUMMARY:
In the case of unitary edentulousness, a dental implant is a prosthetic device fixed in the bone which makes it possible to receive a fixed dental prosthesis (crown). Peri-implant soft tissues (gums) play an essential role in the integration of the crown. Indeed, the implant gingival emergence profile provides an aesthetic integration mimicking that of a natural tooth. This implant emergence profile (EIP) is modeled during the surgical and / or prosthetic phases.

The problem comes from the labile character of the EIP (Emergence Implant Profile). If the literature evokes this problem, the instability of the volume of the EIP during the impression phases has never been measured. Moreover, the three-dimensional behavior of the EIP over time (kinetic) during the acquisition phases is not known.

Objective study of the mobility of gingival tissues of the implant emergence profile (IEP), using an intra-oral optical camera, would scientifically measure the labile aspect of the IEP and improve the procedure of registration of peri-implant soft tissues

DETAILED DESCRIPTION:
Objective study of the mobility of gingival tissues of the implant emergence profile (IEP), using an intra-oral optical camera, would scientifically measure the labile aspect of the IEP and improve the procedure of registration of peri-implant soft tissues.

The main objective is to study the effect of removal of a healing abutment on the closure of the EIP volume at 5 minutes.

This non-interventional study is a prospectively recruited research of the participants and a cross-sectional measure of the judgment criteria (during a single visit). The study is mono-centric, it will take place in the odontology department of Toulouse Hospital.

The question is to know if the decrease in the volume of the PEI is significant during the preparatory phase of the implant impression where the PEI is no longer supported by the healing screw over a period of 5 minutes.

Optical impressions are designed to record adjacent implant site teeth and peri-implant soft tissue PEI using a Optical Camera. The optical camera works like a camera and does not come into contact with the patient's mucous membranes or teeth. The images obtained are saved in STL format on an anonymized file.

ELIGIBILITY:
Inclusion Criteria:

* Patient from the Department of Dentistry who has received an implant in the maxillary or mandible, anterior sector or 1st premolar, and presents himself for the prosthetic stages of the implant treatment (realization of the crown of use),
* Patient affiliated with Social Security,
* Patient having given no objection to his participation in this study
* Good written and oral comprehension of French

Exclusion Criteria:

* Patient who has received an implant intended to receive a removable prosthesis.
* Patient under court bail, tutelage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient from the Department of Dentistry who has received an implant in the maxillary or mandible, anterior sector or 1st premolar, and presents himself for the prosthetic stages of the implant treatment
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Calculation of the volume of the PEI from to T5 min | 5 minutes
  Calculation of the volume of the PEI at T0 min from T5 min :
  They will be named respectively:
  - Flight T0 min : The reference volume is the volume of the PEI at T0 min, it corresponds to the volume of the healing screw created during the mucosal healing phase and which must be kept for the production of the crown of use. It will be called: Vol T0 min. Hypothesis H0 is that Vol T0 min is fixed over time.
  If a volume change of 10% is observed, it is assumed that the clinical consequences are real and that the IEP volume will be undersized compared to the reference IEP. This will have aesthetic and functional consequences.
  The measurement tool of the study is the intraoral scanner.

SECONDARY OUTCOMES:
The volume variation as a percentage of Vol T0.5 min and Vol T2 min | 5 minutes
  The volume variation as a percentage of Vol T0.5 min and Vol T2 min relative to the reference volume Vol T0 min.
The null hypothesis H0 will be a zero variation | 2 years
  The null hypothesis H0 will be a zero variation : a T30 Vol with a Vol T2 min Vol equal to Vol T0 min.
  This Reference Volume is compared to the PEI volume at 5 min: Vol T5 min. If a volume change of 10% is observed, it is assumed that the clinical consequences are real and that the IEP volume will be undersized compared to the reference PEI. This will have aesthetic and functional consequences.
  The reference volume is the volume of the PEI at T0 min, it corresponds to the volume of the healing screw created during the mucosal healing phase and which must be kept for the production of the crown of use. It will be called: Vol T0 min. Hypothesis H0 is that Vol T0 min is fixed over time.
Hypothesis H1 will be a percentage of positive and successively larger variation of Vol T30 dry and Vol T2 min. | 2 years
  Hypothesis H1 will be a percentage of positive and successively larger variation of Vol T30 dry and Vol T2 min.
  This Reference Volume is compared to the PEI volume at 5 min: Vol T5 min. If a volume change of 10% is observed, it is assumed that the clinical consequences are real and that the PEI volume will be undersized compared to the reference PEI. This will have aesthetic and functional consequences.
  The reference volume is the volume of the PEI at T0 min, it corresponds to the volume of the healing screw created during the mucosal healing phase and which must be kept for the production of the crown of use. It will be called: Vol T0 min. Hypothesis H0 is that Vol T0 min is fixed over time.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine GALIBOURG, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No